CLINICAL TRIAL: NCT04523389
Title: Contents of Circulating Extracellular Vesicles: Biomarkers in Colorectal Cancer Patients
Acronym: ExoColon
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: COTTET 2020
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Proteins; Lipids; RNA; Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Non-codant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- colorectal cancer
  Interventions: Biological: analysis (protein, lipid, RNA ...) of circulating exosomes, size and number; Other: Gathering additional information about the patient's cancer; Diagnostic Test: Diagnostic test

INTERVENTIONS:
Biological: analysis (protein, lipid, RNA ...) of circulating exosomes, size and number — use of blood samples stored at the Ferdinand Cabanne Biological Resource Centre
Other: Gathering additional information about the patient's cancer — Gathering additional information about the patient's cancer, its treatment and its sequelae from the patient's medical record.
Diagnostic Test: Diagnostic test — Diagnostic test

SUMMARY:
Most cancer-related deaths are caused by distant metastases, which are tumour cells that have escaped from a primary tumour and passed into the bloodstream to colonize a new organ. In this context, communication between tumour and stromal cells is essential. Indeed, tumor cells interact with cells in the tumor microenvironment and are able to modify them to their advantage. Both extracellular vesicles (EVs) and exosomes are heterogeneous populations of small vesicles present in the tumor microenvironment and in body fluids that have recently emerged as powerful mediators involved in this communication and their transport in fluids. Tumor cells release large quantities of exosomes containing tumor markers, which can then spread to distant locations.

The exosomes are of endosomal origin. They are composed of proteins, lipids, RNA and DNA, and they circulate in the bloodstream. They can be internalized by specific distant cells and thus deliver a functional message. It has recently been shown that tumor exosomes containing pro-metastatic factors form pre-metastatic niches, before the tumor cells actually arrive, while determining the metastatic organotropism of tumors. These properties are now opening up new avenues of research in tumor biomarkers. In recent years, several studies have highlighted different markers contained specifically in exosomes derived from cancer cells. Consequently, exosomes are considered as potential reservoirs of tumor biomarkers that could be clinically useful for the non-invasive diagnosis of cancer, with the advantage of being performed by liquid biopsy. The study of microRNA (miRNA) is of particular interest. Indeed, miRNAs are small non-coding RNAs (between 21 and 25 nucleotides) involved in the regulation of gene expression and which are frequently deregulated in cancer. Several studies underline that the variation of free miRNAs in the blood is correlated with the progression of the disease, particularly in colon cancer. However, the stability of free miRNAs is controversial. Therefore, exosomes represent a very advantageous means of transporting miRNAs in the blood, as they are able to protect miRNAs from degradation by RNAase.

The hypothesis of the project is that circulating exosomes derived from tumours contain markers including specific miRNAs that could be used as biomarkers of early prognosis (survival and progression), easily measured in blood samples from patients with colon cancer. But other molecules contained in exosomes could also be of interest.

ELIGIBILITY:
Inclusion Criteria:

* Person included in the AGARIC study
* Person who provided consent or non-opposition to inclusion in the study
* Available blood sample in the AGARIC biobank at the Biological Resource Centre (Dijon)

Exclusion Criteria:

NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with colorectal cancer and included in the AGARIC study between 2008 and 2012
Sampling Method: Non-Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Prognostic role of exosomes and their contents on the survival of colorectal cancer patients | throughout the study a average of 1 year
  main criterion of judgment: occurrence of death until 30/06/2020
Association between the number and size of exosomes and their content on cancer stage and progression | throughout the study a average of 1 year
  * cancer stage to diagnosis
  * progression of the disease assessed according to the RECIST criteria and defined as (i) local-regional relapse, (ii) distant relapse, (iii) metastasis, (iv) development of another cancer until 30/06/2020.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France